CLINICAL TRIAL: NCT04044885
Title: Investigating the Preferred Nap Schedule for Adolescents With Adequate Sleep
Brief Title: Investigating Preferred Nap Schedules for Adolescents
Acronym: NFS5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Michael WL Chee, MBBS, Principal Investigator, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NFS5
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Sleep
Keywords: Nap; Recovery sleep; Cognitive functions; Neurobehavioural functions; Mood; Subjective sleepiness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nap (Experimental): After each night with a 6.5-hour sleep opportunity, participants have a daytime nap opportunity of 1.5 hours.
  Interventions: Behavioral: Nap
- No nap (No Intervention): After each night with a 8-hour sleep opportunity, participants do not have a daytime nap opportunity, but instead have free time.

INTERVENTIONS:
Behavioral: Nap — Looking at the difference between continuous sleep opportunities and split-sleep opportunities.
  Arms: Nap

SUMMARY:
The aim of this study is to examine the neurobehavioural responses to two successive cycles of sleep manipulation nights and recovery nights in adolescents, and to determine the benefits of napping on cognitive performance, alertness and mood. Using a split-sleep design, 60 participants, aged 15 to 19 years old, are divided into a nap and a no-nap group. Both groups undergo two cycles of sleep manipulation nights and recovery nights over a period of 15 days. The no-nap group receives an 8-hour sleep opportunity on sleep restriction nights, with no daytime nap opportunity. The nap group receives a 6.5-hour sleep opportunity on sleep restriction nights, and has a 1.5-hour nap opportunity the following afternoon.

DETAILED DESCRIPTION:
The present study investigates whether a continuous stretch of night time sleep (8 hours) will lead to better neurobehavioural outcomes relative to nocturnal sleep restriction (6.5 hours) and daytime nap (1.5 hours) of the same total duration. The 15-day protocol is conducted in a dormitory on 60 high school students, aged 15 to 19 years old. Participants are assigned to a nap or no-nap group. Both groups start with two 9-hour adaptation and baseline nights, followed by two successive cycles of sleep restriction (6.5-h time in bed (TIB); 00:15-06:45 or 8-h TIB; 23:30-07:30) and recovery (9-h TIB; 23:00-08:00). Following each sleep-restricted night, the nap group receives a 1.5-h nap opportunity, while participants in the no-nap group watch a documentary. Throughout the protocol, sleep-wake patterns are assessed with actigraphy and polysomnography. Sleepiness levels, mood, vigilance, working memory / executive functions, and speed of processing are assessed 3 times daily (10:00, 16:15, and 20:00).

All participants stay in air-conditioned, twin-share bedrooms with en-suite bathrooms. Bedroom windows are fitted with blackout panels to ensure participants are not woken up prematurely by sunlight. Earplugs are provided, and participants are allowed to adjust the temperature of their bedrooms to their personal comfort. Three main meals are served each day, with snacks being provided for upon request. Caffeinated drinks, unscheduled sleep, and strenuous physical activities are prohibited.

Outside of scheduled sleep, meal, and cognitive testing times, participants spend the majority of their free time in a common room that is illuminated by natural and artificial lighting. They are allowed to read, play non-physically exerting games, watch videos, and interact with research staff and other participants. Participants are under constant supervision by the research staff.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* no sleep disorder
* body mass index not greater than 30

Exclusion Criteria:

* smoker
* habitual short sleeper (time in bed during term time of less than 6 hours and no sign of -
* sleep extension of greater than 1 hour on weekends)
* consumption of more than 5 cups of caffeinated beverages a day
* travelling across more than 2 time zones in the month prior to the study protocol
* diagnosed with any psychiatric conditions

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
1.Change in sustained attention assessed with the Psychomotor Vigilance Task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 16:15, and 20:00) for 15 days
  Number of attention lapses (>500ms)
2.Change in working memory assessed with the 1-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 16:15, and 20:00) for 15 days
  Number of correct responses in the 1-back task
3.Change in executive functions assessed with the 3-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 16:15, and 20:00) for 15 days
  Number of correct responses in the 3-back task
4.Change in the level of subjective sleepiness assessed with the Karolinska Sleepiness Scale from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 16:15, and 20:00) for 15 days
  Score on the Karolinska Sleepiness Scale (1-9 points)
5.Change in positive mood assessed with the Positive and Negative Affect Scale (PANAS) from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 16:15, and 20:00) for 15 days
  Total score on the positive subscale of the PANAS
6.Change in negative mood assessed with the Positive and Negative Affect Scale (PANAS) from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 16:15, and 20:00) for 15 days
  Total score on the negative subscale of the PANAS
7.Change in speed of processing assessed with the Mental Arithmetic Task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 16:15, and 20:00) for 15 days
  Number of correct responses in the task
8.Change in speed of processing assessed with the Symbol Digit Modalities Task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 16:15, and 20:00) for 15 days
  Number of correct responses in the task
11.Change in memory performance in picture-word association task over sleep restriction nights and recovery night | 12 times (morning and evening): after sleep restriction night 1, 2, 3, 4 and 5 (sleep restriction period 1) and after recovery night 2 (recovery period 1)
  Score on picture-word association task
14.Effect of sleep versus wake during delay on memory for rewarded pictures, where the pictures will be encoded either before a 12-hr interval including a night of sleep or a day of wakefulness | Single session during the 15-day protocol, after baseline night 1 or before sleep restriction night 1 (first sleep restriction period)
  Memory score of correctly remembered encoded pictures following the wake or sleep
15.Effect of sleep restriction on learning of novel material (about different animal species) across separate sessions | Single session during the 15-day protocol, after recovery night 2 (first recovery period)
  Memory score on test of learned material
16.Effect of sleep restriction on memory of spatial locations | Single session during the 15-day protocol, after sleep restriction night 3 (first sleep restriction period)
  Performance in four mountains task
18.Effect of sleep restriction on picture encoding | Single session during the 15-day protocol, after recovery night 2 (second recovery period)
  Memory score of correctly remembered encoded pictures of non-famous people, landscapes, scenes and objects
19.Effect of sleep restriction on effort/temporal discounting | Three sessions during the 15-day protocol (after baseline night 1, after sleep restriction night 5 (first sleep restriction period) and after recovery night 2 (first recovery period))
  Choice preference (perform a longer duration task for a higher reward, or to take a break for a lower/no reward) in effort/temporal discounting task is measured

SECONDARY OUTCOMES:
Change in total sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep restriction and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 5 & 7 (first sleep restriction period), 8 (first recovery period), 10 & 12 (second sleep restriction period), & 13 (second recovery period)
  Total duration of nocturnal sleep was determined to establish baseline sleep characteristics (first and second nights) and changes in the first sleep restriction period (third, fifth and seventh night), the first recovery period (eighth night), the second sleep restriction period (tenth and twelfth night), and the second recovery period (13th night).
Change in N1 sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep restriction and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 5 & 7 (first sleep restriction period), 8 (first recovery period), 10 & 12 (second sleep restriction period), & 13 (second recovery period)
  Duration of nocturnal N1 sleep was determined to establish baseline sleep characteristics (first and second nights) and changes in the first sleep restriction period (third, fifth and seventh night), the first recovery period (eighth night), the second sleep restriction period (tenth and twelfth night), and the second recovery period (13th night).
Change in N2 sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep restriction and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 5 & 7 (first sleep restriction period), 8 (first recovery period), 10 & 12 (second sleep restriction period), & 13 (second recovery period)
  Duration of nocturnal N2 sleep was determined to establish baseline sleep characteristics (first and second nights) and changes in the first sleep restriction period (third, fifth and seventh night), the first recovery period (eighth night), the second sleep restriction period (tenth and twelfth night), and the second recovery period (13th night).
Change in N3 sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep restriction and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 5 & 7 (first sleep restriction period), 8 (first recovery period), 10 & 12 (second sleep restriction period), & 13 (second recovery period)
  Duration of nocturnal N3 sleep was determined to establish baseline sleep characteristics (first and second nights) and changes in the first sleep restriction period (third, fifth and seventh night), the first recovery period (eighth night), the second sleep restriction period (tenth and twelfth night), and the second recovery period (13th night).
Change in Rapid Eye Movement (REM) sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep restriction and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 5 & 7 (first sleep restriction period), 8 (first recovery period), 10 & 12 (second sleep restriction period), & 13 (second recovery period)
  Duration of nocturnal REM sleep was determined to establish baseline sleep characteristics (first and second nights) and changes in the first sleep restriction period (third, fifth and seventh night), the first recovery period (eighth night), the second sleep restriction period (tenth and twelfth night), and the second recovery period (13th night).
Change in total sleep duration during daytime naps assessed with polysomnography from the first to the second sleep restriction period | Afternoon naps on days 4, 6 & 8 (first sleep restriction period), 11 & 13 (second sleep restriction period
  Total duration of sleep during the selected nap episodes was determined to track changes in this parameter from the first sleep restriction period (third, fifth and seventh day) to the second sleep restriction period (tenth and twelfth day)
Change in N1 sleep duration during daytime naps assessed with polysomnography from the first to the second sleep restriction period | Afternoon naps on days 4, 6 & 8 (first sleep restriction period), 11 & 13 (second sleep restriction period
  Duration of N1 sleep during the selected nap episodes was determined to track changes in this parameter from the first sleep restriction period (third, fifth and seventh day) to the second sleep restriction period (tenth and twelfth day)
Change in N2 sleep duration during daytime naps assessed with polysomnography from the first to the second sleep restriction period | Afternoon naps on days 4, 6 & 8 (first sleep restriction period), 11 & 13 (second sleep restriction period
  Duration of N2 sleep during the selected nap episodes was determined to track changes in this parameter from the first sleep restriction period (third, fifth and seventh day) to the second sleep restriction period (tenth and twelfth day)
Change in N3 sleep duration during daytime naps assessed with polysomnography from the first to the second sleep restriction period | Afternoon naps on days 4, 6 & 8 (first sleep restriction period), 11 & 13 (second sleep restriction period
  Duration of N3 sleep during the selected nap episodes was determined to track changes in this parameter from the first sleep restriction period (third, fifth and seventh day) to the second sleep restriction period (tenth and twelfth day)
Change in REM sleep duration during daytime naps assessed with polysomnography from the first to the second sleep restriction period | Afternoon naps on days 4, 6 & 8 (first sleep restriction period), 11 & 13 (second sleep restriction period
  Duration of REM sleep during the selected nap episodes was determined to track changes in this parameter from the first sleep restriction period (third, fifth and seventh day) to the second sleep restriction period (tenth and twelfth day)

CONTACTS AND LOCATIONS:
Overall Officials: Michael WL Chee, MBBS, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leong RLF, Tian L, Yu N, Teo TB, Ong JL, Chee MWL. Bidirectional associations between the duration and timing of nocturnal sleep and daytime naps in adolescents differ from weekdays to weekends. Sleep. 2024 Sep 9;47(9):zsae147. doi: 10.1093/sleep/zsae147. PMID 38938171
- [Derived] Golkashani HA, Ghorbani S, Leong RLF, Ong JL, Chee MWL. Advantage conferred by overnight sleep on schema-related memory may last only a day. Sleep Adv. 2023 Apr 14;4(1):zpad019. doi: 10.1093/sleepadvances/zpad019. eCollection 2023. PMID 37193282
- [Derived] Aghayan Golkashani H, Leong RLF, Ghorbani S, Ong JL, Fernandez G, Chee MWL. A sleep schedule incorporating naps benefits the transformation of hierarchical knowledge. Sleep. 2022 Apr 11;45(4):zsac025. doi: 10.1093/sleep/zsac025. PMID 35090173
- [Derived] Lo JC, Koa TB, Ong JL, Gooley JJ, Chee MWL. Staying vigilant during recurrent sleep restriction: dose-response effects of time-in-bed and benefits of daytime napping. Sleep. 2022 Apr 11;45(4):zsac023. doi: 10.1093/sleep/zsac023. PMID 35089345
- [Derived] Leong RLF, Yu N, Ong JL, Ng ASC, Jamaluddin SA, Cousins JN, Chee NIYN, Chee MWL. Memory performance following napping in habitual and non-habitual nappers. Sleep. 2021 Jun 11;44(6):zsaa277. doi: 10.1093/sleep/zsaa277. PMID 33313925
- [Derived] Lo JC, Leong RLF, Ng ASC, Jamaluddin SA, Ong JL, Ghorbani S, Lau T, Chee NIYN, Gooley JJ, Chee MWL. Cognitive effects of split and continuous sleep schedules in adolescents differ according to total sleep opportunity. Sleep. 2020 Dec 14;43(12):zsaa129. doi: 10.1093/sleep/zsaa129. PMID 32619240